CLINICAL TRIAL: NCT07333989
Title: Effect of Biofeedback Activation on Balance in Osteoporotic Elderly Patients
Brief Title: Effect of Biofeedback Activation on Balance in Osteoporotic Elderly
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Said Alsafy Alhamrawy (Other)
Responsible Party: Sponsor-Investigator, Mohamed Said Alsafy Alhamrawy, Doctor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005451
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Balance Problems; Elderly (People Aged 65 or More)
Keywords: Osteoporosis; Elderly; Balance training; Gluteus medius; Electromyography biofeedback; Quality of life; performance.
MeSH Terms: conditions — Osteoporosis | interventions — Electromyography; Biofeedback, Psychology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gluteus medius isometric strengthening using EMG with traditional balance training (Experimental): received 30 minutes of traditional balance training (functional strength, static and dynamic balance, and gait training) followed by 30 minutes of gluteus medius isometric strengthening using EMG biofeedback, three times per week, for four consecutive weeks.
  Interventions: Device: Electromyographic (EMG) biofeedback
- Traditional balance training only (Active Comparator): received balance training alone with the same frequency and duration.
  Interventions: Other: Balance training

INTERVENTIONS:
Device: Electromyographic (EMG) biofeedback — a physical therapy intervention that uses auditory and visual feedback to control the contraction or relaxation of muscles. Repeated biofeedback training can induce motor learning of muscles. Biofeedback enhances the function of pelvic floor muscles by enhancing the force generation, correct timing, and coordination of the pelvic floor muscles. Electromyography Biofeedback is considered as a behavioural therapy training modality
  Arms: Gluteus medius isometric strengthening using EMG with traditional balance training
Other: Balance training — functional strength, static and dynamic balance, and gait training
  Arms: Traditional balance training only

SUMMARY:
This study aimed to investigate the effect of gluteus medius activation using electromyography (EMG) biofeedback combined with balance training on balance, physical performance, gluteus medius muscle activity, and quality of life in osteoporotic elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients included in this study met the following criteria:

  1. Sixty patients of both sexes were diagnosed with osteoporosis confirmed by bone density test through Dual-energy X-ray absorptiometry (DEXA) scan (A T-score equal to or less than - 2.5) (Sheu and Diamond, 2016).
  2. Their age ranged between 65 - 75 years.
  3. Their BMI ranged between 25 - 29.9 kg/m2.
  4. They had good mentality and cognitive function.

Exclusion Criteria:

* The potential patients were excluded if they have one of the following criteria:

  1. Patients with endocrine disorders likely to be related to metabolic bone disease, such as premature ovarian failure, hypogonadism, untreated hyperthyroidism, hyperparathyroidism, adrenal insufficiency or Cushing's syndrome.
  2. Patients with active contagious skin conditions.
  3. Patients with implant devices such as pacemaker or electrical prosthesis.
  4. Any cardiopulmonary disorders.
  5. Any neuromuscular disorders.
  6. Any acute viral infection.
  7. Patients with ascites or end stage liver or kidney failure.
  8. Leg discrepancy.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-04-05 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Balance | Base line before treatment, then one month after treatment
  balance of osteoporotic elderly patients (antero-posterior, medio-lateral, and overall stability indices; Berg Balance Scale)

SECONDARY OUTCOMES:
gluteus medius activity | Base line before treatment and reassessment after one month of treatment
  Assessment of gluteus medius strength by hand-held dynamometer

IPD SHARING:
Plan to Share IPD: No